CLINICAL TRIAL: NCT04703088
Title: A PROSPECTIVE, RANDOMIZED, DOUBLE-BLINDED STUDY OF THE EFFECT OF A STANDARD DOSE OF INTRAVENOUS ONDANSETRON ON THE EFFECTIVE DOSE IN 50% OF SUBJECTS OF PROPHYLACTIC NOREPINEPHRINE INFUSIONS FOR PREVENTING SPINAL ANESTHESIA-INDUCED HYPOTENSION DURING CESAREAN DELIVERY
Brief Title: ONDANSETRON AND EFFECTIVE DOSE IN 50% OF SUBJECTS OF PROPHYLACTIC NOREPINEPHRINE INFUSIONS FOR PREVENTING SPINAL ANESTHESIA-INDUCED HYPOTENSION DURING CESAREAN DELIVERY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laval University (Other)
Collaborators: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Romain LANCHON, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-5610
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Hypotension; Anesthesia; Adverse Effect, Spinal and Epidural; Cesarean Section
Keywords: Spinal Anesthesia; Hypotension, Vascular; Ondansetron Hydrochloride; Norepinephrine; Vasoconstrictor Agents; Cesarean section; Physiological Effects of Drugs; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Hypotension | interventions — Ondansetron; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized blinded parallel assignment
Who Masked: Participant, Care Provider
Masking Description: Studied medication will be administered to the patient after randomization by the investigators (two anesthesia residents or two staff anesthesiologists) who will not be involved in subsequent anesthetic management of the patients. The investigators will also program the infusion rate of norepinephrine at the start of each case and will be the only persons aware of the assigned infusion rate. The investigators will hide the infusion rate with an opaque paper cover over the infusion display during the case.
  The investigators will also collect all the data during each procedures. To summarize, the anesthesiologist in charge of the patient will not know which treatment will be injected and the rate of the pump infusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INTERVENTION GROUP - ONDANSETRON (Experimental): 2 mL of a solution of Ondansetron containing 2mg/ml in a 3 ml syringe will be given intravenously to a patient five minutes before positioning for induction of spinal anesthesia
  Interventions: Drug: Ondansetron 4 MG
- CONTROL GROUP - NORMAL SALINE (Placebo Comparator): 2 mL of 0.9% Saline in a 3 ml syringe will be given intravenously to a patient five minutes before positioning for induction of spinal anesthesia
  Interventions: Drug: 0.9% Saline

INTERVENTIONS:
Drug: Ondansetron 4 MG — 2 mL of a solution of Ondansetron containing 2mg/ml in a 3 ml syringe will be given intravenously to a patient five minutes before positioning for induction of spinal anesthesia
  Arms: INTERVENTION GROUP - ONDANSETRON
Drug: 0.9% Saline — 2 mL of 0,9% Saline in a 3 ml syringe will be given intravenously to a patient five minutes before positioning for induction of spinal anesthesia
  Arms: CONTROL GROUP - NORMAL SALINE

SUMMARY:
Spinal anesthesia is the preferred technique for elective cesarean section as per ASA guidelines. Hypotension is the main complication of this technique and is secondary to both sympatholysis and its associated decrease in systemic vascular resistance and to the Bezold-Jarisch reflex, which causes hypotension and bradycardia in response to noxious stimuli detected in the cardiac ventricles. In pregnant patients, spinal anesthesia induced hypotension is worsened by compression of the aorta and inferior vena cava by the gravid uterus. In this setting, hypotension could lead to uteroplacental hypoperfusion and fetal distress.

In its 2020 guidelines for enhanced recovery after cesarean section, SOAP states that preventing spinal-induced hypotension is an important strategy to enhance maternal and neonatal outcomes in cesarean delivery

Recent studies showed that 5-hydroxytryptamine-3 receptor antagonists, mostly used as nausea and vomiting prophylaxis agents, also contributed to inhibit the Bezold-Jarisch reflex and its associated hemodynamic consequences. Ondansetron is the most studied molecule in this field.

Many recent studies and meta-analyses show renewed interest in the use of norepinephrine as a first line agent for preventing and treating spinal anesthesia-induced hypotension in obstetric anesthesia practice instead of phenylephrine. Norepinephrine has the advantage of a better cardiac output and cardiac frequency as compared to phenylephrine without any fetal side effect. The combination of ondansetron and phenylephrine for the prevention of spinal anesthesia-induced hypotension has been studied, but not the combination of ondansetron and norepinephrine.

The main objective of this study is to evaluate the sparing effect of a standard dose of ondansetron on norepinephrine consumption during elective cesarean section under spinal anesthesia by determining the effective dose in 50% of subjects (ED50) of a prophylactic norepinephrine infusion after receiving a single dose of 4 mg of ondansetron or a saline control.

DETAILED DESCRIPTION:
Vital signs are measured in the preparation area before entrance in the operation theater. The following measures are taken in the supine position every three minutes for three measures: blood pressure and cardiac frequency. The mean blood pressure and cardiac frequency become the reference measure for each patient.

Upon entrance in the operation theater, anesthesia care is given in a standardized manner:

* Supine positioning of the parturient on the operating table
* Standard monitoring of vitals signs every minute for the time of the study, including systolic, diastolic an mean blood pressures, cardiac frequency and SpO2
* 18G intravenous catheter insertion on the forearm
* Randomization of the patient in one of the two groups followed by blind administration of ondansetron or saline
* 5 minute wait period before sitting the patient for spinal anesthesia
* Standardized spinal anesthesia: Whitacre 25G spinal needle, L4-L5 intervertebral space, hyperbaric bupivacaine 12mg + fentanyl 10 mcg + morphine 100 mcg
* Upon injection of the spinal medication: 1000 ml Ringer lactate coloading and start of the iv norepinephrine infusion upon study protocol.
* Evaluation of the sensitive block level at 5 and 10 minutes, a level of T6 is needed to start surgery
* Nausea and vomiting prophylaxis in both groups with metoclopramide 10 mg and dexamethasone 4 mg if no contraindication. Nausea and vomiting per cesarean section will be treated with dimenhydrinate 25 mg
* Bradycardia (HR below 60) will be treated with atropine 0,4 mg
* Multimodal post-operative analgesia with intra rectal acetaminophen 1000 mg and indomethacin 100 mg

Norepinephrine infusion protocol:

* The rate of the infusion pump is blindly set in mcg/kg/min by one of the investigators before the entrance of the patient and the anesthesia team in the operating room. The setting is hidden from the main physician at all times and the perfusion is started when the spinal medication is injected.
* For the first patient of each group (saline and ondansetron) the norepinephrine infusion is started at 0,05 mcg/kg/min until the end of the study
* Hypotension (as defined as a value inferior or equal to 80% of the systolic blood pressure reference value) is treated by the anesthesiologist with a 4 mcg bolus of norepinephrine from a prepared syringe of norepinephrine 4 mcg/ml
* Hypertension (as defined as a value superior or equal to 120% of the systolic blood pressure reference value) is treated by stopping the norephineprine infusion and restarting it when the value is inferior to 120% of the reference value.
* For the following patients, the norepinephrine infusion rate will be adjusted by up and down allocation following the results of the previous patient: if no hypotension occurred (no bolus needed): the infusion rate is decreased by 0,005 mcg/kg/min (for example from 0,05 mcg/kg/min to 0,045 mcg/kg/min) / if at least one hypotension occurred (at least one bolus needed): the infusion rate is increased by 0,005 mcg/kg/min (for example from 0,05 mcg/kg/min to 0,055 mcg/kg/min)

The study is stopped at the fetal delivery.

ELIGIBILITY:
Inclusion Criteria:

* parturients with a singleton pregnancy at term (37 week's gestation and more)
* elective cesarean delivery under spinal anesthesia
* American Society of Anesthesiologists physical status < III

Exclusion Criteria:

* patient refusal
* allergy or hypersensitivity to Norepinephrine or Ondansetron
* Use of monoamine oxidase inhibitors, triptyline or imipramine antidepressants
* Long QT syndrome or another cause of prolonged QT
* significant preexisting maternal disease (cardiovascular or cerebrovascular disease or coagulopathy, diabetes mellitus)
* pre-existing or pregnancy-induced hypertension
* pathological pregnancy (ruptured membranes, pre-eclampsia, placenta praevia, gestational diabetes)
* body mass index < 18 or > 40
* height < 150 or > 180
* fetal abnormalities
* contraindication to spinal anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
ED50 Norepinephrine | At the fetal delivery
  The effective dose in 50% of subjects (ED50) of a prophylactic norepinephrine infusion for preventing hypotension in patients who received a single dose of intravenous ondansetron 4mg or saline control five minutes before spinal anesthesia for elective cesarean delivery

SECONDARY OUTCOMES:
Total consumption of Norepinephrine | At the fetal delivery
  The total consumption of Norepinephrine (mcg/kg) in the two groups (pump infusion and bolus)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Practice Guidelines for Obstetric Anesthesia: An Updated Report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia and the Society for Obstetric Anesthesia and Perinatology. Anesthesiology. 2016 Feb;124(2):270-300. doi: 10.1097/ALN.0000000000000935. No abstract available. PMID 26580836
- [Background] Liu SS, McDonald SB. Current issues in spinal anesthesia. Anesthesiology. 2001 May;94(5):888-906. doi: 10.1097/00000542-200105000-00030. No abstract available. PMID 11388543
- [Background] Klohr S, Roth R, Hofmann T, Rossaint R, Heesen M. Definitions of hypotension after spinal anaesthesia for caesarean section: literature search and application to parturients. Acta Anaesthesiol Scand. 2010 Sep;54(8):909-21. doi: 10.1111/j.1399-6576.2010.02239.x. Epub 2010 Apr 23. PMID 20455872
- [Background] Mercier FJ, Auge M, Hoffmann C, Fischer C, Le Gouez A. Maternal hypotension during spinal anesthesia for caesarean delivery. Minerva Anestesiol. 2013 Jan;79(1):62-73. Epub 2012 Nov 18. PMID 23135692
- [Background] Kinsella SM, Tuckey JP. Perioperative bradycardia and asystole: relationship to vasovagal syncope and the Bezold-Jarisch reflex. Br J Anaesth. 2001 Jun;86(6):859-68. doi: 10.1093/bja/86.6.859. PMID 11573596
- [Background] Malin GL, Morris RK, Khan KS. Strength of association between umbilical cord pH and perinatal and long term outcomes: systematic review and meta-analysis. BMJ. 2010 May 13;340:c1471. doi: 10.1136/bmj.c1471. PMID 20466789
- [Background] Reynolds F, Seed PT. Anaesthesia for Caesarean section and neonatal acid-base status: a meta-analysis. Anaesthesia. 2005 Jul;60(7):636-53. doi: 10.1111/j.1365-2044.2005.04223.x. PMID 15960713
- [Background] Bollag L, Lim G, Sultan P, Habib AS, Landau R, Zakowski M, Tiouririne M, Bhambhani S, Carvalho B. Society for Obstetric Anesthesia and Perinatology: Consensus Statement and Recommendations for Enhanced Recovery After Cesarean. Anesth Analg. 2021 May 1;132(5):1362-1377. doi: 10.1213/ANE.0000000000005257. PMID 33177330
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Fitzgerald JP, Fedoruk KA, Jadin SM, Carvalho B, Halpern SH. Prevention of hypotension after spinal anaesthesia for caesarean section: a systematic review and network meta-analysis of randomised controlled trials. Anaesthesia. 2020 Jan;75(1):109-121. doi: 10.1111/anae.14841. Epub 2019 Sep 18. PMID 31531852
- [Background] Heesen M, Klimek M, Hoeks SE, Rossaint R. Prevention of Spinal Anesthesia-Induced Hypotension During Cesarean Delivery by 5-Hydroxytryptamine-3 Receptor Antagonists: A Systematic Review and Meta-analysis and Meta-regression. Anesth Analg. 2016 Oct;123(4):977-88. doi: 10.1213/ANE.0000000000001511. PMID 27537930
- [Background] Karacaer F, Biricik E, Unal I, Buyukkurt S, Unlugenc H. Does prophylactic ondansetron reduce norepinephrine consumption in patients undergoing cesarean section with spinal anesthesia? J Anesth. 2018 Feb;32(1):90-97. doi: 10.1007/s00540-017-2436-x. Epub 2017 Dec 14. PMID 29243058
- [Background] Gao L, Zheng G, Han J, Wang Y, Zheng J. Effects of prophylactic ondansetron on spinal anesthesia-induced hypotension: a meta-analysis. Int J Obstet Anesth. 2015 Nov;24(4):335-43. doi: 10.1016/j.ijoa.2015.08.012. Epub 2015 Aug 22. PMID 26421701
- [Background] Qian J, Liu L, Zheng X, Xiao F. Does an Earlier or Late Intravenous Injection of Ondansetron Affect the Dose of Phenylephrine Needed to Prevent Spinal-Anesthesia Induced Hypotension in Cesarean Sections? Drug Des Devel Ther. 2020 Jul 16;14:2789-2795. doi: 10.2147/DDDT.S257880. eCollection 2020. PMID 32764878
- [Background] Singh PM, Singh NP, Reschke M, Ngan Kee WD, Palanisamy A, Monks DT. Vasopressor drugs for the prevention and treatment of hypotension during neuraxial anaesthesia for Caesarean delivery: a Bayesian network meta-analysis of fetal and maternal outcomes. Br J Anaesth. 2020 Mar;124(3):e95-e107. doi: 10.1016/j.bja.2019.09.045. Epub 2019 Dec 4. PMID 31810562
- [Background] Heesen M, Hilber N, Rijs K, Rossaint R, Girard T, Mercier FJ, Klimek M. A systematic review of phenylephrine vs. noradrenaline for the management of hypotension associated with neuraxial anaesthesia in women undergoing caesarean section. Anaesthesia. 2020 Jun;75(6):800-808. doi: 10.1111/anae.14976. Epub 2020 Feb 3. PMID 32012226
- [Background] Xu S, Shen X, Liu S, Yang J, Wang X. Efficacy and safety of norepinephrine versus phenylephrine for the management of maternal hypotension during cesarean delivery with spinal anesthesia: A systematic review and meta-analysis. Medicine (Baltimore). 2019 Feb;98(5):e14331. doi: 10.1097/MD.0000000000014331. PMID 30702617
- [Background] Xiao F, Wei C, Chang X, Zhang Y, Xue L, Shen H, Ngan Kee WD, Chen X. A Prospective, Randomized, Double-Blinded Study of the Effect of Intravenous Ondansetron on the Effective Dose in 50% of Subjects of Prophylactic Phenylephrine Infusions for Preventing Spinal Anesthesia-Induced Hypotension During Cesarean Delivery. Anesth Analg. 2020 Aug;131(2):564-569. doi: 10.1213/ANE.0000000000004534. PMID 31725021
- [Background] Ngan Kee WD, Lee SW, Ng FF, Tan PE, Khaw KS. Randomized double-blinded comparison of norepinephrine and phenylephrine for maintenance of blood pressure during spinal anesthesia for cesarean delivery. Anesthesiology. 2015 Apr;122(4):736-45. doi: 10.1097/ALN.0000000000000601. PMID 25635593
- [Background] Ngan Kee WD, Lee SWY, Ng FF, Khaw KS. Prophylactic Norepinephrine Infusion for Preventing Hypotension During Spinal Anesthesia for Cesarean Delivery. Anesth Analg. 2018 Jun;126(6):1989-1994. doi: 10.1213/ANE.0000000000002243. PMID 28678073
- [Background] Sharkey AM, Siddiqui N, Downey K, Ye XY, Guevara J, Carvalho JCA. Comparison of Intermittent Intravenous Boluses of Phenylephrine and Norepinephrine to Prevent and Treat Spinal-Induced Hypotension in Cesarean Deliveries: Randomized Controlled Trial. Anesth Analg. 2019 Nov;129(5):1312-1318. doi: 10.1213/ANE.0000000000003704. PMID 30113395
- [Background] Ngan Kee WD, Lee SWY, Ng FF, Lee A. Norepinephrine or phenylephrine during spinal anaesthesia for Caesarean delivery: a randomised double-blind pragmatic non-inferiority study of neonatal outcome. Br J Anaesth. 2020 Oct;125(4):588-595. doi: 10.1016/j.bja.2020.05.057. Epub 2020 Jul 15. PMID 32682556
- [Background] Wang M, Zhuo L, Wang Q, Shen MK, Yu YY, Yu JJ, Wang ZP. Efficacy of prophylactic intravenous ondansetron on the prevention of hypotension during cesarean delivery: a dose-dependent study. Int J Clin Exp Med. 2014 Dec 15;7(12):5210-6. eCollection 2014. PMID 25664023
- [Background] Pace NL, Stylianou MP. Advances in and limitations of up-and-down methodology: a precis of clinical use, study design, and dose estimation in anesthesia research. Anesthesiology. 2007 Jul;107(1):144-52. doi: 10.1097/01.anes.0000267514.42592.2a. PMID 17585226
- [Background] Dixon, W. J. The Up-and-Down Method for Small Samples. J. Am. Stat. Assoc. (2012).
- [Background] Choi SC. Interval estimation of the LD50 based on an up-and-down experiment. Biometrics. 1990 Jun;46(2):485-92. PMID 2364133
- [Background] Hasanin AM, Amin SM, Agiza NA, Elsayed MK, Refaat S, Hussein HA, Rouk TI, Alrahmany M, Elsayad ME, Elshafaei KA, Refaie A. Norepinephrine Infusion for Preventing Postspinal Anesthesia Hypotension during Cesarean Delivery: A Randomized Dose-finding Trial. Anesthesiology. 2019 Jan;130(1):55-62. doi: 10.1097/ALN.0000000000002483. PMID 30335625
- [Background] Vallejo MC, Attaallah AF, Elzamzamy OM, Cifarelli DT, Phelps AL, Hobbs GR, Shapiro RE, Ranganathan P. An open-label randomized controlled clinical trial for comparison of continuous phenylephrine versus norepinephrine infusion in prevention of spinal hypotension during cesarean delivery. Int J Obstet Anesth. 2017 Feb;29:18-25. doi: 10.1016/j.ijoa.2016.08.005. Epub 2016 Aug 28. PMID 27720613
- [Background] Ngan Kee WD. A Random-allocation Graded Dose-Response Study of Norepinephrine and Phenylephrine for Treating Hypotension during Spinal Anesthesia for Cesarean Delivery. Anesthesiology. 2017 Dec;127(6):934-941. doi: 10.1097/ALN.0000000000001880. PMID 28872480